CLINICAL TRIAL: NCT04797156
Title: The Effect of Combined Intravenous and Topical TXA in Major Multilevel Spine Surgery: A Prospective Randomized Trial
Brief Title: Combined IV and Topical TXA in Major Spine Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Yan Lai, Assistant Professor, Anesthesiology, Perioperative & Pain Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: GCO 19-1137
Record Dates: First submitted 2021-03-10; First posted 2021-03-15 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Spine Surgery; Back Pain
Keywords: tranexamic acid; Spine surgery
MeSH Terms: conditions — Back Pain | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Intervention Model Description: Patients will be assigned randomly using a computer-generated table of numbers to one of the three groups:
  1. High Dose Intravenous TXA (hTXA group)
  2. Low Dose Intravenous TXA (lTXA group)
  3. Combined Intravenous and Topical TXA group (cTXA group).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The patient, surgeon, and anesthesiologist in the case will be blinded
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- High Dose Intravenous TXA (hTXA group) (Experimental): Patients assigned to hTXA group will receive 50mg/kg IV TXA loading dose with a 5mg/kg/hr maintenance dose, and normal saline poured over 5 minutes at the wound prior to closure.
  Interventions: Drug: High Dose Tranexamic acid; Drug: Normal saline
- Low Dose Intravenous TXA (lTXA group) (Experimental): Patients assigned to lTXA group will receive 20mg/kg IV TXA loading dose with a 5mg/kg/hr maintenance dose, and normal saline poured over 5 minutes at the wound prior to closure.
  Interventions: Drug: Low Dose Tranexamic acid; Drug: Normal saline
- Combined Intravenous and Topical TXA group (cTXA group) (Placebo Comparator): Patients assigned to cTXA group will received 20mg/kg V TXA loading dose with a 5mg/kg/hr maintenance dose, and 2g topical TXA poured over 5 minutes at the would prior to closure
  Interventions: Drug: Low Dose Tranexamic acid; Drug: Tranexamic acid Topical

INTERVENTIONS:
Drug: High Dose Tranexamic acid — 50mg/kg IV TXA
  Other Names: hTXA
  Arms: High Dose Intravenous TXA (hTXA group)
Drug: Low Dose Tranexamic acid — 20mg/kg IV TXA
  Other Names: lTXA
  Arms: Combined Intravenous and Topical TXA group (cTXA group); Low Dose Intravenous TXA (lTXA group)
Drug: Tranexamic acid Topical — 2g topical TXA
  Other Names: TXA
  Arms: Combined Intravenous and Topical TXA group (cTXA group)
Drug: Normal saline — Normal saline poured on wound
  Other Names: NS
  Arms: High Dose Intravenous TXA (hTXA group); Low Dose Intravenous TXA (lTXA group)

SUMMARY:
This is a randomized study. The purpose of this study is to evaluate the effect of tranexamic acid in patients undergoing multilevel spine surgery. 75 patients undergoing multi-level spine surgery will be enrolled at Mount Sinai West. Study participation will last from the time of pre-operative evaluation to the time of discharge from hospital. Specifically, the study team will compare tranexamic acid given only intravenously vs. given both topically and intravenously vs. given only intravenously but at a higher dosage. The study team hypothesizes that patient who received combined topical and intravenous TXA (low dose) have similar or decreased overall blood loss postoperatively compared to patient who received high or low dose intravenous TXA alone.

DETAILED DESCRIPTION:
Prospective triple-blinded randomized control trial. The surgeon will provide study information (protocol, consent, general information) to patients in the surgeon's office. Recruitment will be done through a coordination of the operating schedule and the surgeon's office. Patients presenting for preoperative visits at the surgeon's office or the preoperative joint clinic will be approached. On the day of the surgery, the subject will meet the research team in the holding area. The team will finalize participation and ask the subject about the signed consent forms and answer any additional questions. All patients will be provided with copies of the IRB protocol and consent if they wish to have it. Copy of the consent form will be sent in a secured email to the potential subject. The email will be secured by entering in [SECURE] in the e-mail subject line. Once recruited blinding assessments will be done by the study team.

Patients will be assigned randomly using a computer-generated table of numbers to one of the three groups: 1) High Dose Intravenous TXA (hTXA group), 2) Low Dose Intravenous TXA (lTXA group), or 3) Combined Intravenous and Topical TXA group (cTXA group). Surgical team will perform the required spine procedure. Study personnel will make the medication which will be labelled as study drug for surgical and anesthesia team to give during the procedure. Patients assigned to hTXA group will receive 50mg/kg IV TXA loading dose with a 5mg/kg/hr maintenance dose, and normal saline poured over 5 minutes at the wound prior to closure. Patients assigned to lTXA group will receive 20mg/kg IV TXA loading dose with a 5mg/kg/hr maintenance dose, and normal saline poured over 5 minutes at the wound prior to closure. Patients assigned to cTXA group will received 20mg/kg V TXA loading dose with a 5mg/kg/hr maintenance dose, and 2g topical TXA poured over 5 minutes at the would prior to closure. Otherwise, the patient, surgeon, and anesthesiologist in the case will be blinded.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-80 years old
* Undergo major multilevel spine surgery (2-8 levels)
* Male or female

Exclusion Criteria:

* ASA class V
* Urgent or emergent surgery,
* Morbid obesity
* Patients with known coagulopathy disorder, hx of thromboembolic event <1 year, renal insufficiency, hepatic dysfunction, serious cardiac disease
* Patients with known allergy to TXA or receiving antiplatelet and/or anticoagulant drugs
* Religious or other belief that limit blood transfusion,
* Surgery duration more than 6 hours
* Patient refusal or inability to consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Change in Hematocrit level | Baseline and Post-operative day 1, 2 and 3
  The amount of post-operative blood loss during the first 24, 48 and 72 hours in patients undergoing multilevel spine surgery. Specifically, the hematocrit number difference between baseline and post-operative day 1, 2 and 3.

SECONDARY OUTCOMES:
Post-operative drain output | Post-operative day 1, 2 and 3
  The amount of post-operative drain output (ml) during the first 24, 48 and 72 hours in patients undergoing multilevel spine surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Lai, M.D., Principal Investigator — Mount Sinai West and Morningside Hospitals
Locations (1):
- Mount Sinai West Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-10-04): https://cdn.clinicaltrials.gov/large-docs/56/NCT04797156/ICF_000.pdf